CLINICAL TRIAL: NCT04064268
Title: Anabolic Potential of Adding 3-hydroxybutyrate (3-OHB) to Whey Protein in a Catabolic Inflammatory Disease Model: A Human Randomized Controlled Trial
Brief Title: Anabolic Potential of 3-hydroxybutyrate (3-OHB) and Whey Protein in a Human Catabolic Inflammatory Disease Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla Foods Ingredients (Unknown); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Ketone Study
Record Dates: First submitted 2019-07-11; First posted 2019-08-21 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-07

CONDITIONS: Endotoxemia; Muscle Loss; Catabolic State; Protein; Disease; Nutrition Therapy
Keywords: endotoxemia; muscle loss; catabolic state; whey protein; 3-hydroxy butyrate
MeSH Terms: conditions — Endotoxemia; Muscular Atrophy; Disease | interventions — Whey

STUDY DESIGN:
Intervention Model Description: In a randomized crossover design, eight healthy lean young men will undergo either:
  i) Healthy conditions (overnight fast) + whey protein ii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest) + whey protein iii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest) + 3-OHB/whey protein
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy + Whey (Experimental): Healthy conditions (overnight fast)
  Interventions: Dietary Supplement: Whey
- Catabolic + Whey (Experimental): Catabolic conditions (36-hour fast, bed rest and inflammation (LPS))
  Interventions: Dietary Supplement: Whey
- Catabolic + 3-OHB / Whey (Experimental): Catabolic conditions (36-hour fast, bed rest and inflammation (LPS))
  Interventions: Dietary Supplement: 3-OHB + Whey

INTERVENTIONS:
Dietary Supplement: Whey — 45 g whey + 20 g maltodextrin
  Arms: Catabolic + Whey; Healthy + Whey
Dietary Supplement: 3-OHB + Whey — 50 g ketone + 45 g whey + 20 g maltodextrin
  Arms: Catabolic + 3-OHB / Whey

SUMMARY:
This study aims to investigate the muscle anabolic potential of adding ketone (3-hydroxybutyrate) to whey protein compared with isocaloric, isonitrogenous whey protein in a human model of inflammatory catabolic disease. Further, this study aims to investigate whether the same amount of whey protein has different effects on muscles in an catabolic inflammatory setting compared with a healthy setting.

DETAILED DESCRIPTION:
Background: Muscle wasting during hospitalization is caused by a combination of immobilization (bed rest), hypocaloric diet and inflammation (e.g. sepsis), and preventive measures are needed. Whey protein is particularly potent in inducing muscle protein synthesis compared with other proteins, at least in healthy populations. Further, the ketone body 3-hydroxybutyrate (3-OHB) effectively preserved muscle in a model of acute inflammatory disease. However, little is known about whether 3-OHB can potentiate the effects of whey protein in a catabolic inflammatory setting.

Aim: This study aims to investigate the muscle anabolic potential of adding ketone (3-OHB) to whey protein compared with isocaloric, isonitrogenous whey protein in a human model of catabolic inflammatory disease. Further, this study aims to investigate whether the same amount of whey protein has different effects on muscles in an catabolic inflammatory setting compared with a healthy setting.

Hypothesis:

1. 3-OHB potentiates the effect of whey protein in maintaining muscle mass in a catabolic inflammatory setting.
2. The same amount of whey protein will have decreased muscle anabolic effects during catabolic inflammatory conditions compared with healthy conditions

   Interventions:

   In a randomized crossover design, eight healthy, lean, young men will undergo either:

   i) Healthy conditions (overnight fast) + whey protein^ ii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest*) + whey protein^ iii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest*) + 3-OHB/whey protein^"

   *LPS will be administered (1 ng/kg) the day prior to the study together with fast and bed rest. On the study day LPS (0.5 ng/kg) will be injected.

   ^Beverages will be isonitrogenous and isocaloric (fat will be added) with 45 g whey protein + 20 g maltodextrin. Bolus/sip administration will be applied (1/3 bolus, 1/2 sip)

   " 50 grams of 3-OHB will be orally administered (1/2 bolus, 1/2 sip)

   Before each study day:

   The participants arrive fasting (only tap water allowed) by taxi on the study days. They have been without febrile disease the week prior to investigation, and have not performed exercise for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Between 20-40 years of age
* Body mass index between 20-30 kg/m^2
* Healthy
* Oral and written consent forms obtained prior to study day

Exclusion Criteria:

* Recent immobilization of an extremity that is not fully rehabilitated
* Lactose, lidocain or rubber allergies
* Current disease
* Use of anabolic steroids
* Smoking
* Former major abdominal surgery (Or current problems with the GI tract)
* >10 hours of exercise/weak
* Present ketogenic diets or high-protein diets
* Blood doner that does not want to discontinue blood donations until study completion
* Pending MR scan

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Change in forearm muscle kinetics measured by phenylalanine tracer (Netbalance, rate of disappearence and rate of apperance of phenylanine, nmol/100ml muscle/min) | Change from baseline to 3.5 hours after intervention
  Changes of forearm muscle phenylalanine kinetics from baseline to 3.5 hours after intervention using the forearm model

SECONDARY OUTCOMES:
Change in concentration of total aminoacids | Change from baseline to 3.5 hours after intervention
  Change in total aminoacids from baseline to the end of the 3.5 hour sipping period
Change in concentration of 3-hydroxybutyrate (mmol/L) ) | Measured at baseline and every 30. min throughout the 3.5 hour sipping period
  Change in blood BHB levels from baseline to the end of the 3.5 hour sipping period (iAUC)
Change in glucose kinetics measured by glucose tracer (rate of apperance and rate of disappearance, mg/kg/min) | Change from baseline to 3.5 hours after intervention
  Change in glucose kinetics from baseline to to the end of the 3.5 hour sipping period
Change in concentration of plasma insulin | Measured at baseline and every 30. min throughout the 3.5 hour sipping period
  Change in plasma insulin levels from baseline to the end of the 3.5 hour sipping period (iAUC)
Change in concentration of plasma glucose | Measured at baseline and every 30. min throughout the 3.5 hour sipping period
  Change in glucose levels from baseline and after 3.5 hour sipping period expressed as iAUC.
Change in concentration of free fatty acids (FFA) levels | Change from baseline to 3.5 hours after intervention
  Change in FFA from baseline to the end of the sipping period
Change in concentration of C-reactive peptide (CRP) | Change from baseline to 3.5 hours after intervention
  Change in CRP from baseline to the end of the sipping period
Change in concentration of blood leucocytes (x10^9/L) | Change from baseline to 3.5 hours after intervention
  Change in leucocytes from baseline to the end of the sipping period
Change in concentration of stress hormones (glucagon, cortisol, adrenalin, noradrenalin) | Change from baseline to 3.5 hours after intervention
  Change in hormones from baseline and after 3.5 hour sipping period
Change in intracellular muscle signalling | Change from baseline to 3.5 hours after intervention
  Change in muscle signalling in muscle biopsies by western blot from baseline to the sipping period
Difference in muscle forearm kinetics measured by phenylalanine tracer (Netbalance, rate of apperance, rate og disappearance) (healthy vs catabolic) | measured at the end of the 3.5 hour basal period
  Phenylalanine forearm kinetics measured by phenylalanine tracer at the end of the 3.5 hour basal period in healthy vs catabolic (pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure)
Difference in concentration of total amino acids (healthy vs catabolic) | measured at the end of the 3.5 hour basal period
  Total amino acids measured at the end of the 3.5 hour basal period in healthy vs catabolic conditions (pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure)
Difference in glucose kinetics measured with glucose tracer (mg/kg/min) (healthy vs catabolic) | measured at the end of the 3.5 hour basal period
  Glucose kinetics measured by glucose tracer at the end of the 3.5 hour basal period in healthy vs catabolic conditions (pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure)
Difference in concentration of free fatty acids (FFA) (healthy vs catabolic) | Measured at the end of the 3.5 hour basal period.
  FFA measured at the end of the basal period in healthy vs catabolic (pooled mean of the two catabolic days)
Difference in concentration of C-reactive peptide (CRP) (healthy vs catabolic) | Measured at the end of the 3.5 hour basal period.
  CRP measured at the end of the basal period in healthy vs catabolic (pooled mean of the two catabolic days)
Difference in concentration of leucocytes (healthy vs catabolic) | Measured at the end of the 3.5 hour basal period.
  Leucocytes measured at the end of the basal period in healthy vs catabolic (pooled mean of the two catabolic days)
Difference in intracellular muscle signalling (healthy vs catabolic) | Measured at the end of the 3.5 hour basal period.
  Muscle signalling measured in muscle biopsies by western blot during the 3.5 hour basal period in healthy vs catabolic (pooled mean of the two catabolic days)
Difference in concentration of 3-hydroxybutyrate (mmol/L) (healthy vs catabolic) | Measured at the end of the 3.5 hour basal period.
  3-hydroxybutyrate measured at the end of the basal period in healthy vs catabolic (pooled mean of the two catabolic days)
Difference in concentration of hormones (insulin, glucagon, cortisol, growth hormone, adrenaline, noradrenalin) (healthy vs catabolic) | Measured at the end of the 3.5 hour basal period.
  Hormones (insulin, glucagon, cortisol, growth hormone, adrenaline, noradrenalin) measured at the end of the basal period in healthy vs catabolic (pooled mean of the two catabolic days)
Difference in whole body protein metabolism (healthy vs catabolic) | Measured at the end of the 3.5 hour basal period.
  Difference in whole body protein metabolism measured with tyrosine tracers at the end of the basal period in healthy vs catabolic (pooled mean of the two catabolic days)
Difference in concentration of cytokines (healthy vs catabolic) | Measured at baseline and 120 and 240 minutes after LPS administration
  Cytokines (TNFalfa, IL-10, IL-6 and IL-1beta) measured between healthy and catabolic conditions (iAUC, a pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure))
Difference in axillary temperature (healthy vs catabolic) | Measured at baseline and 1, 2, 3, 4, 5, 6 and 7 hours after LPS administration
  Change in axillary temperature (iAUC). A pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure.
Difference in heart rate (healthy vs catabolic) | Measured at baseline and 1, 2, 3, 4, 5, 6 and 7 hours after LPS administration
  Change in heart rate (iAUC). A pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure.
Difference in mean arterial pressure (MAP) (healthy vs catabolic) | Measured at baseline and 1, 2, 3, 4, 5, 6 and 7 hours after LPS administration
  Change in MAP (iAUC). A pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure.
Difference in symptom score (healthy vs catabolic) | Measured at baseline and 1, 2, 3, 4, 5, 6 and 7 hours after LPS administration
  Change from baseline and throughout the experiment (iAUC). A pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure. Scale 0-5, 0=no symptoms and 5=severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Niels Moeller, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Medical Research Laboratory, DoH, Aarhus University Hospital, Aarhus, Denmark